CLINICAL TRIAL: NCT05747625
Title: Study Evaluating 89Zr Panitumumab for Assessment of Indeterminate Metastatic Lesions on 18F-FDG-PET/CT in Head and Neck Squamous Cell Carcinoma
Brief Title: (89Zr Panitumumab) With PET/CT for Diagnosing Metastases in Patients With Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eben Rosenthal (Other)
Collaborators: Vanderbilt-Ingram Cancer Center (Other); Vanderbilt University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Barry and Amy Baker Professor and Chair, Vanderbilt-Ingram Cancer Center
Organization: Vanderbilt-Ingram Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: VICCHN2279; NCI-2023-01365 (Registry Identifier: NCI, Clinical Trials Reporting Program)
Record Dates: First submitted 2023-02-16; First posted 2023-02-28 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Stage IV Cutaneous Squamous Cell Carcinoma of the Head and Neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Panitumumab; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (89Zr panitumumab PET/CT) (Experimental): Patients receive panitumumab IV, 89Zr panitumumab IV, and undergo PET/CT on study
  Interventions: Biological: Panitumumab; Drug: Zirconium Zr 89 Panitumumab; Procedure: Positron Emission Tomography; Procedure: Computed Tomography; Other: Electronic Health Record Review

INTERVENTIONS:
Biological: Panitumumab — Given IV
Drug: Zirconium Zr 89 Panitumumab — Given IV
Procedure: Positron Emission Tomography — Undergo PET/CT
Procedure: Computed Tomography — Undergo PET/CT
Other: Electronic Health Record Review — Ancillary studies

SUMMARY:
The goal of this phase I clinical trial is to evaluate the usefulness of an imaging test (zirconium Zr89 panitumumab [89Zr panitumumab]) with positron emission tomography (PET)/computed tomography (CT) for diagnosing the spread of disease from where it first started (primary site) to other places in the body (metastasis) in patients with head and neck squamous cell carcinoma. Traditional PET/CT has a low positive predictive value for diagnosing metastatic disease in head and neck cancer. 89Zr panitumumab is an investigational imaging agent that contains radiolabeled anti-EGFR antibody which is overexpressed in head and neck cancer. The main question this study aims to answer is the sensitivity and specificity of 89Zr panitumumab for the detection of indeterminate metastatic lesions in head and neck cancer.

Participants will receive 89Zr panitumumab infusion and undergo 89Zr panitumumab PET/CT 1 to 5 days after infusion. Participants will otherwise receive standard of care evaluation and treatment for their indeterminate lesions.

Researchers will compare the 89Zr panitumumab to standard of care imaging modalities (magnetic resonance imaging (MRI), CT, and/or PET/CT).

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

- Determine the sensitivity and specificity of zirconium Zr 89 panitumumab (89Zrpanitumumab) for the detection of indeterminate metastatic lesions in head and neck squamous cell carcinoma.

SECONDARY OBJECTIVE:

- Compare sensitivity and specificity of standard of care imaging modalities (magnetic resonance imaging [MRI], CT and/or fludeoxyglucose F-18 [18F]-PET/CT) to 89Zr-panitumumab-PET/CT for detection of indeterminate metastatic lesions in head and neck squamous cell carcinoma.

EXPLORATORY OBJECTIVE:

- Determine rate of intervention (e.g., biopsy or other invasive procedures) versus (vs) non-intervention (e.g., serial imaging, observation) by treatment team in subjects with indeterminate metastatic lesions on standard of care imaging.

OUTLINE:

Patients receive panitumumab intravenously (IV), 89Zr panitumumab IV, and undergo PET/CT on study.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 19 years
* Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck
* Subjects diagnosed with any T stage, any subsite within the head and neck. Subjects with recurrent disease or a new primary will be allowed
* Must have evidence of indeterminate metastatic squamous cell carcinoma (SCC) based on 18F-fluorodeoxyglucose (FDG)-PET/CT or Primary SCC with suspicious Lymph Nodes on CT prior to surgical removal
* Hemoglobin >= 9gm/dL
* White blood cell count > 3000/mm^3
* Platelet count >= 100,000/mm^3
* Serum creatinine =< 1.5 times upper reference range

Exclusion Criteria:

* Myocardial infarction (MI); cerebrovascular accident (CVA); uncontrolled congestive heart failure (CHF); significant liver disease; or unstable angina within 6 months prior to enrollment
* History of infusion reactions to other monoclonal antibody therapies
* Pregnant (based on screening serum pregnancy test and day 0 urine pregnancy test administered before unlabeled panitumumab), or breastfeeding
* Magnesium or potassium lower than the normal institutional values
* Subjects receiving class IA (quinidine, procainamide) or class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents
* Subjects with a history or evidence of interstitial pneumonitis or pulmonary fibrosis
* Severe renal disease or anuria
* Known hypersensitivity to deferoxamine or any of its components

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of zirconium Zr 89 panitumumab (89Zr-panitumumab | Up to 7 years
  The total number of head and neck squamous cell carcinoma lesions accurately detected by 89Zr-panitumumab using positron emission tomography (PET)/computed tomography (CT) imaging (test) will be compared with lesions identified as positive during the 36 +/- 6 month follow-up period (gold standard). Significance will be assessed at an alpha level of 0.05 and, to assess uncertainty, 95% confidence intervals will be provided for all estimates.
Specificity of 89Zr-panitumumab | Up to 7 years
  The total number of head and neck squamous cell carcinoma lesions accurately detected by 89Zr-panitumumab using PET/CT imaging (test) will be compared with lesions identified as positive during the 36 +/- 6 month follow-up period (gold standard). Significance will be assessed at an alpha level of 0.05 and, to assess uncertainty, 95% confidence intervals will be provided for all estimates.

SECONDARY OUTCOMES:
Sensitivity of 89Zr-panitumumab | Up to 7 years
  The sensitivity of 89Zr-panitumumab will be compared to the sensitivity of standard of care imaging modalities, including magnetic resonance imaging (MRI), CT, and/or fludeoxyglucose F-18 (18F-FDG) PET/CT. Will use the matched pair Durkalski's test, accounting for the cluster-correlation within subjects, for the sensitivity comparisons.
Specificity of 89Zr-panitumumab | Up to 7 years
  The specificity of 89Zr-panitumumab will be compared to the specificity of standard of care imaging modalities, including MRI, CT, and/or 18F-FDG PET/CT. Will use the matched pair Durkalski's test, accounting for the cluster-correlation within subjects, for the specificity comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Topf, MD, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Informed Consent Form (2025-08-01): https://cdn.clinicaltrials.gov/large-docs/25/NCT05747625/ICF_001.pdf